CLINICAL TRIAL: NCT00241735
Title: Soy Food and Coronary Heart Disease in Women
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1311; R01HL079123 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To investigate whether soy food intake reduces risk of non-fatal myocardial infarction (MI) and fatal coronary heart disease in Chinese women.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD) is the leading cause of death in the US and many other countries. Estrogen deficiency plays a significant role in the development of coronary heart disease (CHD) in postmenopausal women. Recently, a series of randomized clinical trials evaluating the effects of hormone replacement therapy (HRT) on CHD yielded surprisingly deleterious results, shifting clinical decision-making from a position of presumed benefit to one of potential harm. Soy food is emerging as a promising natural substitute for HRT, given its estrogenic properties and potential lipids benefits. However, data directly linking soy food intake to the clinical endpoints of CHD are lacking.

DESIGN NARRATIVE:

The study will evaluate the association of soy food consumption with CHD using resources from the Shanghai Women's Health Study (SWHS), an ongoing prospective cohort study of 75,000 Chinese women who were recruited from 1997 to 2000 and who completed two extensive dietary assessments at baseline. The investigators will verify all CHD events identified in this cohort during the follow-up and longitudinally analyze the association between soy food intake and CHD risk, overall, and according to conventional CHD risk factors. In addition, they will conduct a nested case-control study to evaluate the association of urinary isoflavonoids (a biomarker of soy intake) and risk of CHD, and to investigate whether soy and CHD associations are modified by baseline levels of lipids and plasma C-reactive protein, two well established risk markers of CHD. In the United States, the sale of soy products has increased more than 3-fold in recent decades, and the proportion of people reporting soy product consumption at least once a week nearly doubled in the last six years. However, the overall intake level of soy food in the US population is still low, and women who consume soy food regularly are likely to be highly selective. Furthermore, it is difficult, if at all possible, to assess usual soy food intake in the US population because soy protein is added to many American food products. Informative studies on the association between soy food intake and CHD risk are better conducted in Chinese and other Asian populations, where soy food is part of traditional dietary practice. The SWHS with its wealth of data on dietary and lifestyle factors and biological samples provides a unique and unparalleled opportunity to prospectively investigate the effects of soy food intake on the risk of CHD, and to identify those most likely to benefit from consumption of soy food.

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 135896 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Shu, Principal Investigator — Vanderbilt University Medical Center